CLINICAL TRIAL: NCT00773877
Title: Comparison of RNFL Thickness Measurements by Time-Domain and Spectral-Domain OCT In Glaucoma Patients
Brief Title: Comparison of Retinal Nerve Fiber Layer (RNFL) Thickness Measurements by Time-Domain and Spectral-Domain OCT In Glaucoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Kim Chan Yun, Institute of Vision Research, Department of Ophthalmology, Severance Hospital, Yonsei University School of Medicine
Other Study IDs: 4-2008-0342
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Primary Open Angle Glaucoma
Keywords: RNFL thickness
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Primary open angle glaucoma
- 2: Normal Controls

SUMMARY:
Measurement of RNFL thickness by OCT is at a cornerstone for the correct diagnosis and monitoring of progression of glaucomatous optic neuropathy.

Spectral domain technology has enabled better reproducibility with better axial resolution in the measurement of RNFL thickness. A comparative study among Stratus, Cirrus and RT-View will enable clinicians to determine differences among various instruments.

ELIGIBILITY:
Exclusion Criteria:

* Evidence of retinal disease
* Secondary glaucoma due to intraocular inflammation
* Lens induced glaucoma
* Neovascular glaucoma
* Tumor induced glaucoma

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary open angle glaucoma
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
RNFL thickness | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Severance Hospital, Yonsei University School of Medicine, Seoul, South Korea